CLINICAL TRIAL: NCT02695108
Title: Scapular Stabilization Exercise on Mechanical Neck Pain: A Randomized Control
Brief Title: Scapular Stabilization Exercise on Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Taha İbrahim Yıldız, Research Asistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/498
Record Dates: First submitted 2016-02-09; First posted 2016-03-01 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Neck Pain
Keywords: Scapula; Neck; Pain; Therapy; Kinematic
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- classical approach for neck pain (Experimental): patients in this arm received classical approaches for neck pain. Cervical manual therapy was performed on patients in this arm and they were also instructed to to perform cervical endurance, strength and stretching exercises. Rehabilitation period was lasted for 6 weeks. Pain, quality of life and scapular kinematics were assessed before and after rehabilitation program.
  Interventions: Other: classical approach for neck pain
- scapular exercise on neck pain (Experimental): patients in this arm received cervical manual therapy and cervical exercises too. Apart from cervical manual therapy and cervical exercises,patients also performed scapular stabilization exercise targeting trapezius, serratus anterior and rhomboid muscles. Rehabilitation period was lasted for 6 weeks. The same assessment parameters was conducted on this arm too.
  Interventions: Other: scapular exercise on neck pain

INTERVENTIONS:
Other: classical approach for neck pain — Patients with mechanical neck pain were instructed to do cervical exercise
  Arms: classical approach for neck pain
Other: scapular exercise on neck pain — Patients with mechanical neck pain were instructed to do scapular stabilization and cervical exercise
  Arms: scapular exercise on neck pain

SUMMARY:
Neck pain is a very common problem in the population. Most of the patients suffer from neck pain for long time and the problem becomes chronic. The investigators studied the effects of scapular stabilization exercise on mechanical neck pain.

DETAILED DESCRIPTION:
Neck is one of the most common musculoskeletal problem in the world. Yet the problem still haven't been understood and solved completely. Its incidence is also becoming higher and most people who have neck pain suffer from it for long time. Several problems have been related to neck pain. Hence, the investigators designed a study to see the effects of scapular stabilization exercise on neck pain.

ELIGIBILITY:
Inclusion Criteria:

* having neck pain at least 6 months
* having score of at least 10 points from Neck Disability Index
* having type-1, type-2 or type-3 scapula from Kibler's four types rating system
* no previous shoulder or neck surgery
* no accompanying shoulder problem

Exclusion Criteria:

* no complying to the rehabilitation
* if patient wants to finished and don't want to complete study, they were excluded

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Neck pain measured with Visual Analog Scale | 6 weeks
  Patient's neck was measured with Visual Analog Scale

SECONDARY OUTCOMES:
Quality of Life measured with Neck Disability Index | 6 weeks
  Patient's quality of life was measured with Neck Disability Index
Scapular Kinematics measured with 3-D motion monitor device | 6 weeks
  Patient's scapular kinematics was measured with 3-D motion monitor device

CONTACTS AND LOCATIONS:
Overall Officials: İrem Düzgün, Study Director — supervisor of the study
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Helgadottir H, Kristjansson E, Mottram S, Karduna AR, Jonsson H Jr. Altered scapular orientation during arm elevation in patients with insidious onset neck pain and whiplash-associated disorder. J Orthop Sports Phys Ther. 2010 Dec;40(12):784-91. doi: 10.2519/jospt.2010.3405. Epub 2010 Oct 22. PMID 20972341
- [Result] Helgadottir H, Kristjansson E, Einarsson E, Karduna A, Jonsson H Jr. Altered activity of the serratus anterior during unilateral arm elevation in patients with cervical disorders. J Electromyogr Kinesiol. 2011 Dec;21(6):947-53. doi: 10.1016/j.jelekin.2011.07.007. Epub 2011 Sep 1. PMID 21889362
- [Result] Cagnie B, Struyf F, Cools A, Castelein B, Danneels L, O'leary S. The relevance of scapular dysfunction in neck pain: a brief commentary. J Orthop Sports Phys Ther. 2014 Jun;44(6):435-9. doi: 10.2519/jospt.2014.5038. Epub 2014 May 10. PMID 24816504